CLINICAL TRIAL: NCT03760640
Title: Evaluation of LY900014 in a Medtronic Pump
Brief Title: A Study of LY900014 in a Medtronic Pump
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16917; I8B-MC-ITSM (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Results first posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2019-10-15

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY900014 (Experimental): Participants received 100 units per milliliter (U/mL) of LY900014 administered via continuous subcutaneous insulin infusion (CSII) by the Medtronic MiniMed 670G insulin pump.
  Interventions: Drug: LY900014
- Insulin Lispro (Humalog) (Active Comparator): Participants received 100 U/mL of Insulin lispro (Humalog) administered via CSII by the Medtronic MiniMed 670G insulin pump.
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro; Lyumjev
  Arms: LY900014
Drug: Insulin Lispro — Administered SC
  Other Names: Humalog; LY275585
  Arms: Insulin Lispro (Humalog)

SUMMARY:
The purpose of this study is to compare the study drug LY900014 to insulin lispro (Humalog) when both are delivered by the Medtronic MiniMed 670G System in adults with type 1 diabetes (T1D). The study will consist of two treatment periods of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been diagnosed with type 1 diabetes and have been using insulin continuously for at least 12 months
* Participants must be using an insulin pump with "rapid-acting insulin" for at least 6 months and the same "rapid acting insulin" for at least the past 30 days
* Participants must have hemoglobin A1c (HbA1c) values ≥6.0% and ≤8.0%
* Participants must have been using the MiniMed 670G insulin pump for at least the past 90 days
* Participants must use their Guardian (3) sensor at least an average of 75% of the time and remain in Auto Mode an average of 70% of the time

Exclusion Criteria:

* Participants must not have had more than 1 emergency treatment for very low blood glucose or any hospitalizations for poor glucose control (very high blood sugar or diabetic ketoacidosis) in the last 6 months
* Participants must not have significant abnormal accumulation of fat, loss of fat tissue, or scars just under the skin in areas of infusion or have a history of an infection at an infusion site within 90 days prior to screening
* Participants must not have a total daily insulin dose >100 units
* Participants must not be receiving any oral or injectable medication intended for the treatment of diabetes other than rapid-acting analog insulin via CSII in the 30 days prior to screening
* Participants must not have major problems with their heart, kidneys, liver, or have a blood disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - International Diabetes Center, Saint Louis Park, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Bode B, Carlson A, Liu R, Hardy T, Bergenstal R, Boyd J, Morrett S, Ignaut D. Ultrarapid Lispro Demonstrates Similar Time in Target Range to Lispro with a Hybrid Closed-Loop System. Diabetes Technol Ther. 2021 Dec;23(12):828-836. doi: 10.1089/dia.2021.0184. Epub 2021 Oct 26. PMID 34270335

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Participants received 100 units per milliliter (U/mL) of LY900014 or Insulin lispro delivered via continuous subcutaneous insulin infusion (CSII) using the Medtronic MiniMed 670G insulin pump.
  Period 1: LY900014 Period 2: Insulin Lispro (Humalog)
- Sequence 2: Participants received 100 U/mL of LY900014 or Insulin lispro delivered via CSII using the Medtronic MiniMed 670G insulin pump.
  Period 1: Insulin Lispro (Humalog) Period 2: LY900014
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 20 | 22
Received at Least 1 Dose of Study Drug | 20 | 22
Completed | 20 | 22
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2
Started | 20 | 22
Completed | 20 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Sequence 1: Participants received 100 units per milliliter (U/mL) of LY900014 or Humalog delivered via continuous subcutaneous insulin infusion (CSII) using the Medtronic MiniMed 670G insulin pump.
  Period 1: LY900014 Period 2: Humalog
- Sequence 2: Participants received 100 U/mL of LY900014 or Humalog delivered via CSII using the Medtronic MiniMed 670G insulin pump.
  Period 1: Humalog Period 2: LY900014
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (14.9) | 48.1 (13.1) | 47.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 22 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time With Sensor Glucose Values Between 70 and 180 Milligrams Per Deciliter (mg/dL) (24-Hour)
Description: Least Square (LS) mean was determined by mixed-model repeated measures (MMRM) with baseline, period, sequence, strata (Hemoglobin A1c (HbA1c) [<=7.0%, >7.0%] and percentage of time with sensor glucose values from 70 to 180 mg/dL over the 2 weeks prior to randomization [<=75%, >75%]), treatment (Type III sum of squares) as fixed factors.
Time Frame: Week 2 through Week 4
Population: All randomized participants who received at least one dose of study drug and had at least one post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Time
Groups:
- LY900014: Participants received 100 U/mL of LY900014 delivered via CSII using the Medtronic MiniMed 670G insulin pump.
- Insulin Lispro (Humalog): Participants received 100 U/mL of Insulin lispro delivered via CSII using the Medtronic MiniMed 670G insulin pump.
Arm/Group | LY900014 | Insulin Lispro (Humalog)
Number analyzed (Participants) | 42 | 42
Percentage of Time | 76.98 (0.857) | 77.84 (0.857)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog); Test type: Superiority; p = 0.339, Mixed Models Analysis; LS Mean Difference = -0.86, 90% CI 2-sided [-2.35 to 0.63]

2. Secondary Outcome: Mean Sensor Glucose Value (24-Hour)
Description: LS mean was determined by MMRM with baseline, period, sequence, strata (HbA1c [<=7.0%, >7.0%] and percentage of time with sensor glucose values from 70 to 180 mg/dL over the 2 weeks prior to randomization [<=75%, >75%]), treatment (Type III sum of squares) as fixed factors.
Time Frame: Week 2 through Week 4
Population: All randomized participants who received at least one dose of study drug and had at least one post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY900014 | Insulin Lispro (Humalog)
Number analyzed (Participants) | 42 | 42
milligrams per deciliter (mg/dL) | 148.64 (1.193) | 145.64 (1.193)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog); Test type: Superiority; p = 0.011, Mixed Models Analysis; LS Mean Difference = 3.00, 90% CI 2-sided [1.10 to 4.90]

3. Secondary Outcome: Percentage of Time Spent in Auto Mode
Description: as for outcome 2
Time Frame: Week 2 through Week 4
Population: All randomized participants who received at least one dose of study drug and had at least post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Time
Arm/Group | LY900014 | Insulin Lispro (Humalog)
Number analyzed (Participants) | 42 | 41
Percentage of Time | 91.98 (0.829) | 91.42 (0.838)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog); Test type: Superiority; p = 0.557, Mixed Models Analysis; LS Mean Difference = 0.56, 90% CI 2-sided [-1.02 to 2.14]

4. Secondary Outcome: Percentage of Time With Sensor Glucose Values <54 mg/dL (24-Hour)
Description: as for outcome 2
Time Frame: Week 2 through Week 4
Population: All randomized participants who received at least one dose of study drug and had at least one post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Time
Arm/Group | LY900014 | Insulin Lispro (Humalog)
Number analyzed (Participants) | 42 | 42
Percentage of Time | 0.34 (0.067) | 0.38 (0.067)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog); Test type: Superiority; p = 0.548, Mixed Models Analysis; LS Mean Difference = -0.04, 90% CI 2-sided [-0.15 to 0.07]

5. Secondary Outcome: Rate of Severe Hypoglycemic Events
Description: Severe hypoglycemic is defined as an event requiring assistance of another person to administer carbohydrate, glucagon, or other resuscitative actions. During these episodes, the participant has an altered mental status and cannot assist in his or her own care, or may be semiconscious or unconscious, or experience coma with or without seizures, and may require parenteral therapy. Rate of severe hypoglycemia events per 100 years during a defined period was calculated by total number of severe hypoglycemia episodes within the period divided by the cumulative days on treatment from all participants within a treatment group *36525. No severe hypoglycemia was reported for this study.
Time Frame: Week 2 through Week 4
Population: All randomized participants with evaluable hypoglycemic data.
Measure: Mean (Standard Deviation); unit: Events/Participant/100 Years
Arm/Group | LY900014 | Insulin Lispro (Humalog)
Number analyzed (Participants) | 42 | 42
Events/Participant/100 Years | 0 (0) | 0 (0)

6. Secondary Outcome: Total Daily Insulin Dose
Description: as for outcome 2
Time Frame: Week 2 through Week 4
Population: All randomized participants who received at least one dose of study drug and had at least one post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: Units (U)/day
Arm/Group | LY900014 | Insulin Lispro (Humalog)
Number analyzed (Participants) | 42 | 42
Units (U)/day | 42.59 (1.023) | 42.10 (1.023)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog); Test type: Superiority; p = 0.577, Mixed Models Analysis; LS Mean Difference = 0.49, 90% CI 2-sided [-0.97 to 1.94]

ADVERSE EVENTS:
Time Frame: Up To 10 Weeks
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | LY900014 | Insulin Lispro (Humalog)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 4/42 | 1/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014 (N=42) | Insulin Lispro (Humalog) (N=42)
Infusion site pain (General disorders) | 4 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-04-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT03760640/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT03760640/SAP_001.pdf